CLINICAL TRIAL: NCT06662344
Title: A Randomly Controlled Study to Explore the Effect of Oral Tube Feeding on Sleep Quality in Stroke-related Dysphagia
Brief Title: Nutrition Tubes on Sleep Quality in Stroke-related Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babujinaya Cela (Other Government)
Responsible Party: Sponsor-Investigator, Babujinaya Cela, The Research Director, Buraidah Central Hospital
Organization: Buraidah Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IOE-Sleep
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oral-esophageal Tube Feeding+comprehensive rehabilitation therapy (Experimental): During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on the patients; health condition. The observation group receives Intermittent Oro-esophageal Tube Feeding for enteral nutrition support
  Interventions: Behavioral: Intermittent Oral-esophageal Tube Feeding; Behavioral: comprehensive rehabilitation therapy
- Nasogastric Tube Feeding+comprehensive rehabilitation therapy (Active Comparator): During the 15-day treatment, both groups of patients are hospitalized, while conventional care and enteral nutrition support are provided to the two groups. Specifically, conventional care includes health education, dietary adjustments, nasopharyngeal hygiene, management of risk factors (blood pressure and lipid control, etc.), exercise rehabilitation, and psychological support. The frequency and content of these interventions are arranged based on the patients; health condition.The control group receives nasogastric tube for enteral nutrition support
  Interventions: Behavioral: Nasogastric Tube Feeding; Behavioral: comprehensive rehabilitation therapy

INTERVENTIONS:
Behavioral: Intermittent Oral-esophageal Tube Feeding — The specific procedure was as follows: the infant was placed in a semi-recumbent or sitting position with the head fixed. Before each feeding, the infant's oral and nasal secretions were to be cleared. An intermittent oro-esophageal tube was appropriately lubricated with water on the head part. The professional medical staff held the tube and slowly inserted it through one side of the mouth into the upper part of the esophagus. The depth of insertion depended on the patient's age and height. After each feeding, the tube was immediately removed, and the patient was held upright for at least 30 minutes in case of reflux.
  Arms: Intermittent Oral-esophageal Tube Feeding+comprehensive rehabilitation therapy
Behavioral: Nasogastric Tube Feeding — Nasogastric Tube Feeding were used for feeding to provide nutritional support. Each feeding was administered by a nurse using the infant's mother's breast milk through the tube. The amount of each feeding varied from 20 to 100 ml depending on the age of the infant, with feedings given every 2 to 3 hours, approximately 10 times per day. The duration of each feeding procedure ranged from 10 to 20 minutes. The total daily intake ranged from 200 to 1000 ml. Each tube was kept indwelling for 5 to 7 days. When the tube needed to be replaced, it was removed after the last feeding of a day and a new tube was to be inserted through the other nostril on the following morning to continue the nutritional support.
  Arms: Nasogastric Tube Feeding+comprehensive rehabilitation therapy
Behavioral: comprehensive rehabilitation therapy — Both groups were given comprehensive rehabilitation therapy. The main intervention measures included: 1) non-invasive ventilator treatment, generally at least once every night and typically not exceeding continuous daily usage.; 2) attention to feeding and sleeping positions, with a recommended sleeping position of lateral recumbent and the head of the bed raised by 20-30°; 3) swallowing function training, such as tongue muscle stretching training, assisted anterior jaw protrusion training, lemon ice stimulation to the soft palate, pharyngeal wall, etc., generally 5 days per week, twice per day, 5-20 minutes each time; 4) pulmonary ultrashort wave therapy, generally at least 2-3 times a week, and not more than once a day; 5) physical therapy, such as intensive training for gross motor functions including lifting the head, turning over, sitting, crawling, standing, etc., generally 3-5 days per week, 1-2 times per day, 5-20 min each time.

SUMMARY:
Palliation to stroke-related dysphagia continues to be a challenge. Although nasogastric tube feeding (NGT) has been adopted widely, the weaknesses have yet to be improved by another enteral nutrition support mode.

This study aims to observe the clinical efficacy of intermittent oro-esophageal tube feeding (IOE) in the treatment of stroke-related dysphagia on sleep quality. This is a prospective study with patients with dysphagia after stroke. Patients enrolled are randomly divided equally into 2 groups. All patients receive conventional care, and the observation group received IOE while the control group received NGT for enteral nutrition support.

Their sleep quality are compared at baseline and after study.

DETAILED DESCRIPTION:
This study lasts 15 days for each patient. Palliation to stroke-related dysphagia continues to be a challenge. Although nasogastric tube feeding (NGT) has been adopted widely, the weaknesses have yet to be improved by another enteral nutrition support mode.

This study aims to observe the clinical efficacy of intermittent oro-esophageal tube feeding (IOE) in the treatment of stroke-related dysphagia on sleep quality. This is a prospective study with patients with dysphagia after stroke. Patients enrolled are randomly divided equally into 2 groups. All patients receive conventional care, and the observation group received IOE while the control group received NGT for enteral nutrition support.

Their sleep quality are compared at baseline and after study.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke .
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* No history of prior stroke.
* Stable vital signs.

Exclusion Criteria:

* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | day1 and day15
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used questionnaire that assesses sleep quality and disturbances over a one-month period. It consists of 19 items that are grouped into seven components. Each component is scored from 0 to 3, with a total PSQI score ranging from 0 to 21. A higher score indicates worse sleep quality, while a lower score indicates better sleep quality. Generally, a total score of 5 or higher is considered indicative of poor sleep quality.